CLINICAL TRIAL: NCT01885286
Title: Simple Circumcision Device: Proof-of-Concept for a Single-visit, Adjustable Device to Facilitate Safe Adult Male Circumcision
Brief Title: Pilot Trial of Novel Circumcision Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, John Krieger, Professor of Urology, University of Washington, Section chief Seattle VA urology division, VA Puget Sound Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAPSHCS-00434
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Safe Circumcision
Keywords: circumcision; HIV prevention
MeSH Terms: interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: circumcision with simple circumcision device — Circumcision performed with the device in the operating room using local anesthesia

SUMMARY:
The investigators are testing a novel surgical device to facilitate safe circumcision among adult males. The investigators hypothesize that this device will allow non-medical providers to perform safe surgical circumcision without adverse events.

DETAILED DESCRIPTION:
Objective: To conduct a proof-of-concept study to determine the potential utility of a novel, adjustable single-visit, disposable device to facilitate rapid adult circumcision.

Design: Prospective pilot trial of a novel surgical device Setting: Tertiary care Veterans Administration medical center Patients: 5 adult males Interventions: Circumcisions performed by junior trainees using an adjustable, single-size surgical-assist device constructed by the University of Washington Applied Physics Laboratory.

Main Outcome Measure(s): The attending surgeon and trainees completed standardized forms after each procedure to assess technical problems and ease of use. Follow-up visits were scheduled to evaluate adverse events, post-operative pain, cosmetic outcomes and participant satisfaction at 3, 8, 30 and 90 days post-operatively.

ELIGIBILITY:
Inclusion

1. Uncircumcised males
2. Aged>18
3. Sexually active
4. No plans for moving in next 6 months
5. Consent to participate

Exclusion

1. History of a bleeding disorder
2. History of a documented concurrent STI of appearance of an STI on initial physical exam
3. Keloid formation or other condition that might unduly increase risk of elective surgery
4. Asprin, anti-coagulants or other clinical contra-indications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Efficacy, injury rate, conversion to standard method rate and cosmetic outcomes of novel surgical device | 90 days
  To determine if the novel surgical device was able to facilitate safe circumcision among adult males. Specifically we looked at: time of surgery, blood loss, ease of use, cosmetic outcome, number of sutures required, need for conversion to another method of circumcision and need for revision surgeries.

SECONDARY OUTCOMES:
Time of circumcision | 1 day
  To determine how long the operative procedure required to complete

CONTACTS AND LOCATIONS:
Overall Officials: John N Krieger, MD, Principal Investigator — University of Washington/Seattle Puget Sound VA Health Care System; James M Hotaling, MD MS, Study Director — University of Washington
Locations (1):
- Veterans Administration Puget Sound Health Care System, Seattle, Washington, United States